CLINICAL TRIAL: NCT06919822
Title: SCAN Electrical Stimulation for Idiopathic Parkinson's Disease: A Prospective Open-Label Clinical Trial
Brief Title: SCAN Electrical Stimulation for Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changping Laboratory (Other)
Collaborators: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SES-PD
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Personalized ESE Intervention Arm (Experimental): This experimental arm involves a comprehensive two-stage therapeutic intervention for Parkinson's disease patients:
  * Pre-surgical Screening Stage:
    * All participants first undergo non-invasive intermittent theta-burst stimulation (iTBS) targeting their individualized Somato-Cognitive Action Network (SCAN) region.
  * Surgical Intervention Stage (for iTBS responders):
    * Patients showing ≥30% improvement in motor symptoms proceed to epidural implantation of electrodes over the predetermined SCAN target.
  Interventions: Device: Personalized SCAN Electrical Stimulation

INTERVENTIONS:
Device: Personalized SCAN Electrical Stimulation — * Stage 1: iTBS Intervention (14 days) and Washout Period (3-6 months)
    * All enrolled participants undergo:
      * Baseline clinical assessments
      * Structural and functional MRI with pBFS mapping
      * Resting motor threshold determination
    * Daily iTBS sessions targeting individualized SCAN coordinates:
      * Treatment duration: 14 consecutive days
      * Post-intervention evaluation at Day 14-21
    * Mandatory observation window:
      * No neuromodulation therapies permitted
      * Stable PD medication regimen maintained
      * Monthly safety monitoring
  * Stage 2: Surgical Intervention and Follow-up (12 months)
    * Surgical Procedure:
      * Epidural electrode implantation
      * 7-day externalized stimulation testing
      * Pulse generator internalization
    * Chronic Stimulation Stage:
      * Parameter optimization visits
      * Scheduled follow-ups at Months 1, 3, 6, 9, 12

SUMMARY:
The goal of this clinical trial is to learn if electrical stimulation targeting the Somato-Cognitive Action Network (SCAN) can improve motor symptoms in adults with idiopathic Parkinson's disease (PD). It will also evaluate the safety of this treatment. The main questions it aims to answer are:

* Does electrical stimulation targeting SCAN reduce motor symptoms (measured by MDS-UPDRS-III scores) in PD patients after 3 months?
* Is SCAN electrical simulation (SES) a safe and tolerable treatment for PD, with minimal adverse effects?

Researchers will compare participants' baseline motor function to their post-treatment results to determine if SES is effective.

Participants will:

* First undergo non-invasive brain stimulation (iTBS) to test responsiveness.
* If eligible, receive surgical implantation of SES electrodes in the personalized SCAN target.
* Complete follow-up visits for 12 months to monitor symptoms, side effects, and quality of life.

DETAILED DESCRIPTION:
Background:

This is a prospective, open-label, single-center clinical trial investigating the efficacy and safety of personalized electrical stimulation targeting the Somato-Cognitive Action Network (SCAN) in patients with idiopathic Parkinson's disease (PD). The study employs a two-stage intervention approach with comprehensive clinical and functional assessments. The study builds upon recent discoveries that the SCAN network shows preferential connectivity with PD-affected subcortical structures. By combining advanced neuroimaging for personalized target identification with staged therapeutic intervention, the trial aims to establish proof-of-concept for this novel neuromodulation approach. The design allows for initial non-invasive validation of target engagement through iTBS before proceeding to surgical implantation.

Study Design and Methodology:

The trial consists of two sequential stages:

- Screening and iTBS Intervention Stage (14 days) and a Washout Period (3-6 months): Eligible participants will first undergo intermittent theta-burst stimulation (iTBS) to their individualized SCAN target, identified through resting-state functional MRI and personalized-Brain-Functional-Sector (pBFS) mapping.

Participants demonstrating ≥30% improvement in motor symptoms proceed to a mandatory washout period.

Complete cessation of all neuromodulation therapies while maintaining stable PD medications.

- Surgical Intervention and Follow-up (12 months): Responsive patients undergo epidural electrode implantation over their predetermined SCAN target.

Includes 1-week externalized testing before pulse generator internalization. A scheduled12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with idiopathic Parkinson's disease (PD) according to the revised clinical diagnostic criteria of the International Movement Disorder Society (MDS) (2015 version) or the Chinese Parkinson's Disease Diagnostic Criteria (2016 version).
* Age between 40 and 75 years, with a minimum age of 40 years at the time of diagnosis.
* Any gender, including both male and female patients.
* Hoehn-Yahr staging between 2 and 4 (inclusive).
* Disease duration of 4 years or more.
* Responding effectively to levodopa-based drug therapy with a minimum of 30% improvement in the levodopa loading test.
* Presence of motor fluctuations with or without anisocoria despite optimal drug treatment.
* Stable on medication for at least the past 1 month prior to screening and surgery.
* Ability to understand the trial and willingness to sign an informed consent form.

Exclusion Criteria:

* Diagnosis of Parkinsonian superimposed syndrome or secondary Parkinson's disease.
* Presence of intracranial structural variants or other abnormalities that may interfere with TMS or surgical treatment, as detected by MRI or CT.
* Implantation of metallic medical devices such as deep brain stimulators, cochlear implants, vagus nerve stimulators, etc., which may affect MRI examination and TMS treatment.
* Contraindications to MRI scanning, including claustrophobia, tattoos, or magnetic metal-containing implants (to be confirmed with specialists).
* History of comorbid epilepsy or having first-degree relatives with a history of epilepsy.
* Receipt of other neuromodulation treatments (e.g., TMS, transcranial electrical stimulation, transcranial ultrasound stimulation) within the 3 months prior to enrollment.
* Contraindications to neurosurgery, such as bleeding or coagulation disorders.
* Presence of severe organic diseases, including heart failure, renal failure, or malignancies.
* Cognitive impairment as indicated by MMSE score of 24 or below.
* Significant speech impairment, hearing impairment, or visual impairment that limits cooperation with testing.
* Severe depression (HAMD-17 score of 24 or above) or severe anxiety (HAMA score of 29 or above).
* Diagnosed psychiatric disorders based on DSM-V criteria or any psychological issues that may interfere with the study protocol.
* Alcohol or substance abuse.
* Active infections including hepatitis B virus (HBV), hepatitis C virus (HCV), syphilis, or human immunodeficiency virus (HIV) infection as determined by the investigator.
* Any other medical abnormalities deemed by the investigator to be unsuitable for participation in the trial.
* Inability to complete follow-up visits due to geographical or other reasons.
* Women of childbearing age who are pregnant, breastfeeding, or intend to become pregnant during the trial.
* Participation in other clinical trials concurrently.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in Movement Disorder Society-Unified Parkinson's Disease Rating Scale Part III motor scores at 3 months post-stimulation（medication "off" state） | Baseline to 3 months post-stimulation
  The change in Movement Disorder Society-Unified Parkinson's Disease Rating Scale Part III (MDS-UPDRS-III) motor examination scores measured during the medication "off" state (after 12-hour overnight withdrawal of anti-Parkinson medications) from baseline to 3 months after initiating motor cortex stimulation. Higher scores indicate more severe motor impairment (range 0-132). A negative change indicates improvement.

SECONDARY OUTCOMES:
Change in MDS-UPDRS-III scores (ON/OFF states) from baseline to 12 months | Baseline, 1-week, 1/3/6/9/12 months post-stimulation
  Difference in Movement Disorder Society-Unified Parkinson's Disease Rating Scale Part III (MDS-UPDRS-III) motor examination scores (range 0-132, higher=worse) between baseline and post-stimulation assessments during both medication ON (2 hours after levodopa dose) and OFF (after 12-hour withdrawal) states.
Change in daily OFF time duration (hours) from baseline | Baseline, 1/3/6/9/12 months post-stimulation
  Reduction in self-reported daily hours of OFF periods (time when Parkinson's medications are ineffective) as recorded in patient diaries, comparing baseline to post-stimulation timepoints.
Change in daily ON time duration (hours) without dyskinesia | Baseline, 1/3/6/9/12 months post-stimulation
  Increase in self-reported daily hours of good ON periods (medication effectiveness without troublesome dyskinesia) from baseline to follow-up assessments.
Change in 39-item Parkinson's Disease Questionnaire summary index score from baseline | Baseline, 1/3/6/9/12 months post-stimulation
  Difference in 39-item Parkinson's Disease Questionnaire (PDQ-39) total score (range 0-100, higher=worse quality of life) between baseline and follow-up assessments.
Change in Clinical Global Impression (CGI) score from baseline | Baseline, 1/3/6/9/12 months post-stimulation
  Improvement in clinician-rated CGI scale (range 1-7, higher=worse) assessing overall disease severity change since baseline.
Change in levodopa equivalent daily dose (LEDD) from baseline | Baseline, 3/6/9/12 months post-stimulation
  Reduction in calculated total daily dopaminergic medication dosage (mg/day) while maintaining symptom control.

OTHER OUTCOMES:
Change in Movement Disorder Society-Unified Parkinson's Disease Rating Scale Part I (MDS-UPDRS-I) scores from baseline | Baseline, 1/3/6/9/12 months post-stimulation
  Difference in MDS-UPDRS-I non-motor experiences of daily living scores (range 0-52, higher=worse) between baseline and post-stimulation assessments.
Change in Movement Disorder Society-Unified Parkinson's Disease Rating Scale Part II (MDS-UPDRS-I) scores from baseline | Baseline, 1/3/6/9/12 months post-stimulation
  Difference in MDS-UPDRS-II non-motor experiences of daily living scores (range 0-52, higher=worse) between baseline and post-stimulation assessments.
Change in Movement Disorder Society-Unified Parkinson's Disease Rating Scale Part IV (MDS-UPDRS-I) scores from baseline | Baseline, 1/3/6/9/12 months post-stimulation
  Difference in MDS-UPDRS-IV motor complications scores (range 0-24, higher=worse) assessing dyskinesia and motor fluctuations.
Change in Non-Motor Symptoms Scale (NMSS) score from baseline | Baseline, 1/3/6/9/12 months post-stimulation
  Difference in Non-Motor Symptoms Scale total score (range 0-360, higher=worse) evaluating frequency and severity of non-motor symptoms in Parkinson's disease.
Change in Pittsburgh Sleep Quality Index (PSQI) score from baseline | Baseline, 1/3/6/9/12 months post-stimulation
  Difference in Pittsburgh Sleep Quality Index global score (range 0-21, higher=worse sleep quality) assessing sleep disturbances and patterns.
Change in Hamilton Depression Rating Scale-17 (HAMD-17) score from baseline | Baseline, 1/3/6/9/12 months post-stimulation
  Difference in 17-item Hamilton Depression Rating Scale scores (range 0-52, higher=more severe depression) evaluating depressive symptoms.
Change in Hamilton Anxiety Rating Scale (HAMA) score from baseline | Baseline, 1/3/6/9/12 months post-stimulation
  Difference in Hamilton Anxiety Rating Scale scores (range 0-56, higher=more severe anxiety) assessing anxiety symptoms.
Change in Mini-Mental State Examination (MMSE) score from baseline | Baseline, 3/12 months post-stimulation
  Difference in Mini-Mental State Examination total score (range 0-30, higher=better cognitive function) assessing global cognitive status.
Change in Montreal Cognitive Assessment (MoCA) score from baseline | Baseline, 3/12 months post-stimulation
  Difference in Montreal Cognitive Assessment total score (range 0-30, higher=better cognitive function) evaluating multiple cognitive domains.

CONTACTS AND LOCATIONS:
Overall Officials: Hesheng Liu, PhD, Study Chair — Changping Laboratory
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality, China